CLINICAL TRIAL: NCT05546385
Title: A Prospective, Multi-centre, Randomized, Double-blind, Sham-controlled, Parallel-group, Group-sequential Study to Investigate Safety and Effectiveness of the Rehaler Partial Rebreathing Device, in Adults Suffering From Migraine With Aura
Brief Title: PArtial REbreathing for Migraine With Aura 1
Acronym: PAREMA1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis lack-of-effect stopping condition was met
Sponsor: Rehaler (Industry)
Collaborators: Qmed Consulting A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-001
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, randomized, double-blind, sham-controlled, parallel-group, group-sequential study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active device (Active Comparator)
  Interventions: Device: Partial Rebreathing Device
- Sham device (Placebo Comparator)
  Interventions: Device: Sham breathing device

INTERVENTIONS:
Device: Partial Rebreathing Device — Partial Rebreathing Device
  Arms: Active device
Device: Sham breathing device — Sham breathing device
  Arms: Sham device

SUMMARY:
A prospective, multi-centre, randomized, double-blind, sham-controlled, parallel-group, group-sequential study to investigate safety and effectiveness of the Rehaler partial rebreathing device, in adults suffering from migraine with aura

ELIGIBILITY:
Inclusion Criteria:

1. Participant has migraine with typical aura (ICHD3 classification 1.2.1) with the additional criterion that historically in more than 75% of cases of aura a moderate or severe headache begins between 10 and 60 minutes after aura onset.
2. Participant has had 3 or more migraine-with-aura attacks over the last six months.
3. Participant is 18 to 65 years of age.
4. Participant's age at onset of migraine with aura was less than 50 years.
5. If participant is taking migraine prophylactic drugs, the dose must have been stable for three months or more.
6. Participant agrees to withhold usual acute migraine medications until at least two hours after treatment with the study device.
7. Participant does not plan to initiate new (and/or change existing) migraine prophylaxis medication for the duration of Stage 1 of the study.
8. For female participants: is willing to use adequate contraception during study participation
9. Participant owns a smartphone compatible with the ePRO study diary app.
10. Participant agrees to use the study device as intended, comply with all study requirements including treatment, follow-up visits, and recording required study data in the ePRO app.
11. Participant is willing and able to provide written informed consent.

Exclusion Criteria:

1. Participant has a history of chronic pulmonary disease (e.g. Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis).
2. Participant has a history of severe cardiovascular disease (e.g. symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure) or cerebrovascular disease (e.g. prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery).
3. Participant has a history of intracranial hyper/hypo-tension.
4. Participant has a history of cerebral aneurysm.
5. Participant has had previous brain surgery, including stenting.
6. Anaemia, defined as a hemoglobin concentration in capillary blood lower than 11g/dL
7. Participant has a baseline SPO2 level which is lower than 95% performed at Site Visit 1.
8. Participant has 15 or more headache days per month
9. Participant has medication-overuse headache (ICHD3 classification 8.2).
10. Participant has a known history or suspicion of recurring secondary headache which in the opinion of the investigator may interfere with the study.
11. Hemiplegic migraine
12. Participant has other significant and relevant pain problem (e.g. cancer pain, fibromyalgia or other head or facial pain disorders)
13. Participant has a known history or suspicion of substance abuse or addiction (within the last 5 years) that in the opinion of the investigator may confound the study assessments.
14. Participant has a history of psychiatric or cognitive disorder and/or behavioural problems which in the opinion of the investigator may interfere with the study.
15. Participant belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised (e.g. homeless, developmentally disabled, prisoner).
16. For female participants: is pregnant or actively trying to become pregnant.
17. Participant is participating in any other clinical investigation or has participated in an interventional clinical trial in the preceding 30 days.
18. Participant has any condition that according to the investigator may pose the participant at risk or provide confounding data.
19. Participant is unable, as perceived by study personnel, to correctly understand and follow the instructions for use of the device and ePRO app.
20. Sickle Cell Disease
21. Participant is being treated with nerve blocks or injections for migraine prophylaxis on a regularly scheduled basis (including Botox, Aimovig/Erenumab, Ajovy/Fremanezumab, Emgality/Galcanezumab or Vyepti/Eptinezumab).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (9):
  - Stanford University - Stanford Headache Clinic, Palo Alto, California
  - Profound Research-Southern California Neurology Consultants, Pasadena, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Yale University, New Haven, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - PharmaSite Research, Baltimore, Maryland
  - Clinvest Research, Springfield, Missouri
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Germany (6):
  - Charité University Hospital, Berlin
  - Essen University Hospital-West German Headache Center, Essen
  - Frankfurt Headache Center, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - Jena University Hospital, Jena
  - Munich University Hospital, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gaul C, Ferreira S, Johansen T. Partial rebreathing is not effective for early treatment of migraine with aura attacks: Results of a double-blind, randomized, controlled trial (PAREMA1). Headache. 2025 Nov 21. doi: 10.1111/head.15090. Online ahead of print. PMID 41272403

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Device | Sham Device
Started | 72 | 70
Completed | 13 | 15
Not Completed | 59 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Device | Sham Device | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 70 | 142
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.10 (10.32) | 40.31 (11.38) | 39.19 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 55 | 117
  Male | 10 | 15 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 4 | 7
  Black/African-American | 7 | 6 | 13
  Hispanic/Latino | 6 | 4 | 10
  White/Caucasian | 53 | 54 | 107
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
  Germany | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Absence of Moderate or Severe Pain at 2 Hours (AMSP2)
Description: The percentage of attacks in which the participant reported absence of headache of moderate or severe intensity at 2 hours post-treatment initiation
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 60.0 | 69.7

2. Secondary Outcome: Pain Freedom at 2 Hours (PF2)
Description: The percentage of attacks with absence of headache pain two hours after treatment initiation
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 21.4 | 18.2

3. Secondary Outcome: Freedom From Most Bothersome Symptom at 2 Hours (MBSF2)
Description: The percentage of attacks with absence of MBS two hours after treatment initiation
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 37.1 | 39.7

4. Secondary Outcome: Sustained Pain Freedom at 24 Hours (SPF24)
Description: The percentage of attacks having no headache pain at 2 hours after treatment initiation, with no use of rescue medication and no relapse of headache pain within 24 hours
Time Frame: 24 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 16.7 | 15.9

5. Secondary Outcome: Headache Score at 2 Hours (HS2)
Description: Headache Score 2 hours after treatment initiation. Measured on Likert four-point scale: 0 = no headache; 1 = mild headache; 2 = moderate headache; 3 = severe headache.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 1.29 (0.92) | 1.21 (0.85)

6. Secondary Outcome: Most Bothersome Symptom Score at 2 Hours (MBS2).
Description: Most Bothersome Symptom score two hours after treatment initiation. Measured on Likert four-point scale: 0 = symptom absent; 1 = mild degree of symptom; 2 = moderate degree of symptom; 3 = severe degree of symptom.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 0.87 (0.83) | 0.95 (0.99)

7. Secondary Outcome: Functional Disability Score at 2 Hours (FDS2)
Description: Functional Disability Score two hours after treatment initiation. Measured on Likert four-point scale: 0 = no functional disability; 1 = mild functional disability; 2 = moderate functional disability; 3 = severe functional disability.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 0.77 (0.87) | 0.88 (1.06)

8. Secondary Outcome: Attacks With Use of Rescue Medication From the 2 Hours' Time Point Until 24 Hours (Res24)
Description: The percentage of attacks with use of rescue medication from the 2 hours' time point until 24 hours (Res24)
Time Frame: 24 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 53.7 | 34.4

9. Secondary Outcome: Participant Satisfaction at 48 Hours (PS48)
Description: Participant's overall satisfaction with the acute treatment effect on attack, evaluated at 48 hours after treatment initiation (5 point satisfaction scale: 5 = Satisfied, 4 = Partially Satisfied, 3 = Neutral, 2 = Partially Unsatisfied, 1 = Unsatisfied)
Time Frame: 48 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 3.72 (1.17) | 3.65 (1.14)

10. Secondary Outcome: Light Sensitivity Score at 2 Hours (LSS2)
Description: Photophobia (light sensitivity) score two hours after treatment initiation. Measured on Likert four-point scale: 0 = no photophobia; 1 = mild photophobia; 2 = moderate photophobia; 3 = severe photophobia.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 0.89 (0.83) | 0.86 (0.97)

11. Secondary Outcome: Nausea Score at 2 Hours (NS2)
Description: Nausea Score two hours after treatment initiation. Measured on Likert four-point scale: 0 = no nausea; 1 = mild nausea; 2 = moderate nausea; 3 = severe nausea.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 0.36 (0.57) | 0.56 (0.86)

12. Secondary Outcome: Sound Sensitivity Score at 2 Hours (SSS2)
Description: Phonophobia (sound sensitivity) score two hours after treatment initiation. Measured on Likert four-point scale: 0 = no phonophobia; 1 = mild phonophobia; 2 = moderate phonophobia; 3 = severe phonophobia.
Time Frame: 2 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
score on a scale | 0.64 (0.82) | 0.64 (0.82)

13. Secondary Outcome: Freedom From Relapse at 48 Hours (FR48)
Description: The percentage of attacks having no headache pain at 2 hours after dose, with no use of rescue medication and no relapse of headache pain within 48 hours
Time Frame: 48 hours
Population: Each participant could report more than one attack. In the study, 67 participants reported a total of 136 attacks.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Number of attacks
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 34 | 33
Number analyzed (Number of attacks) | 70 | 66
percentage of attacks | 10.2 | 16.1

ADVERSE EVENTS:
Time Frame: Variable between patients according to their enrolment date (earliest enrolled patients had longer period to report data than latest enrolled patients). Patient with longest duration of period for collecting adverse event = 449 days. Patient with shortest duration of period for collecting adverse event = 14 days.
Arm/Group | Active Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/70
Other Adverse Events (participants affected / at risk) | 2/72 | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Device (N=72) | Sham Device (N=70)
Heavy salivation (General disorders) | 0 (0) | 1 (1) — Sham device
Heavy breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT05546385/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05546385/SAP_001.pdf